CLINICAL TRIAL: NCT01277055
Title: MRI Perfusion Imaging at 3T With TX Parallel RF Technology to Identify Myocardial Ischemia Compared to Invasive FFR Measurements
Brief Title: MRI Perfusion Imaging at 3Tx Compared to Invasive FFR Measurements
Acronym: Vision MRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heart Center Bogenhausen (Other)
Responsible Party: Alexander Leber, MD, Heart Center Bogenhausen
Other Study IDs: HCB10071
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Perfusion Imaging; MRI; Myocardial Fractional Flow Reserve; Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Coronary artery disease (CAD) has a great significance concerning prevalence and mortality in the western world. It is usually diagnosed by catheterization and coronary arteries are visually assessed by the examiner. Thus having a great spectrum of interobserver differences, especially when it comes to intermediate lesions. The gold standard to assess the haemodynamic significance is the measurement of the myocardial fractional flow reserve (FFR). The FAME-study (Tonino, De Bruyne et al. 2009) was able o show that additional FFR- measurements in patients with intermediate lesions could significantly reduce stent implementation and consequently mortality. However this method is not used in daily routine and is available only in a fraction of catheter labs worldwide. Taking this into account decision finding especially in intermediate lesions remains difficult.

One major step to simplify the invasive approach concerning intermediate lesions would be to establish a non-invasive procedures which localizes the coronary vessel to intervene ahead catheterization.

Do to steady technical development cardiac MRI has become a powerful tool which is able to determine myocardial vitality, perfusion and function. In particular the new generation of 3 Tesla multi transmit MR with its higher field strength and better spatial resolution seems to be able to show first pass myocardial perfusion more precise. With this new technology prefixed to cardiac catheterization clinical relevant information can be made accessible and thus reduce the number of unnecessary implemented stents.

ELIGIBILITY:
Inclusion Criteria:

* intermediate lesion defined by myocardial fractional flow reserve measurement
* age > 18 years

Exclusion Criteria:

* pregnancy
* contraindication with adenosin, contrast agents or MR-Scaning
* severe renal dysfunktion
* instable patient(e.g. acute myocardial infarction)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with intermediate lesion who underwent cardiac catheterization inluding measurement of the myocardial fractional flow reserve
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-01

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Center Bogenhausen, Munich Municipal Hospital Group, Munich, Bavaria, Germany